CLINICAL TRIAL: NCT04269629
Title: The Effect of Antihypertensive Drugs on Severity of Anaphylaxis and Side-effects During Venom Immunotherapy
Acronym: EADOAS
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 26-422 ex13/14 (EADOAS)
Record Dates: First submitted 2020-02-05; First posted 2020-02-17 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Hymenoptera Venom Allergy; Antihypertensive Treatment
MeSH Terms: interventions — Arthropod Venoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with a history of an anaphylactic sting reaction: At Visit 1, patients will be included after carefully reviewing all inclusion and exclusion criteria. All data concerning the index sting, laboratory parameters like immunoglobulin E (IgE) and tryptase levels and skin test results will be recorded as well as the concomitant diseases and medication. Visit 2 will be performed after VIT updosing is finished. At this Visit data concerning the immunotherapy - premedication, preparation, updosing protocol, the outcome of possible large, local reactions (LLR) and systemic reactions (SR) and changes in diseases and medication will be recorded. One year after reaching the maintenance dose, Visit 3 will be performed. At this Visit data concerning the maintenance phase like premedication and possible side effects will be recorded as well as the outcome of insect stings.
  Interventions: Drug: Insect Venom

INTERVENTIONS:
Drug: Insect Venom — Patients receive insect venom immunotherapy. The frequency of systemic side-effects is recorded and compared between patients under antihypertensive treatment and patients not taking antihypertensive drugs.

SUMMARY:
There is an ongoing debate whether antihypertensive treatment with beta-blockers and/or angiotensin converting Enzyme (ACE)-inhibitors comprises a risk factor for more severe and more frequent side-effects during venom immunotherapy (VIT). In the literature, data are controversial and originate from case reports or statistically underpowered studies; the number of included patients was usually high but the proportion of patients on antihypertensive treatment was low ranging from 2-11%.

The study was conducted as a prospective, observational, European multicenter study. 1425 patients, aged from 35 to 85 years, with a history of an anaphylactic reaction due to bee or wasp stings, were included. The medical history was recorded as well as laboratory parameters and data of the VIT-updosing phase. One year after reaching the maintenance dose, possible side-effects during VIT as well as the outcome of field stings or sting challenges were documented.

ELIGIBILITY:
Inclusion Criteria:

* History of systemic sting reaction (≥ grade I according the classification by Ring and Messmer)
* age 35 to 85 years

Exclusion Criteria:

* absolute contraindications for VIT
* pretreatment with Omalizumab

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a history of anaphylactic sting reaction
Sampling Method: Probability Sample
Enrollment: 1425 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology and Venerology, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sturm GJ, Herzog SA, Aberer W, Alfaya Arias T, Antolin-Amerigo D, Bonadonna P, Boni E, Bozek A, Chelminska M, Ernst B, Frelih N, Gawlik R, Gelincik A, Hawranek T, Hoetzenecker W, Jimenez Blanco A, Kita K, Kendirlinan R, Kosnik M, Laipold K, Lang R, Marchi F, Mauro M, Nittner-Marszalska M, Poziomkowska-Gesicka I, Pravettoni V, Preziosi D, Quercia O, Reider N, Rosiek-Biegus M, Ruiz-Leon B, Schrautzer C, Serrano P, Sin A, Sin BA, Stoevesandt J, Trautmann A, Vachova M, Arzt-Gradwohl L. beta-blockers and ACE inhibitors are not a risk factor for severe systemic sting reactions and adverse events during venom immunotherapy. Allergy. 2021 Jul;76(7):2166-2176. doi: 10.1111/all.14785. Epub 2021 Mar 11. PMID 33605465

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With a History of an Anaphylactic Sting Reaction: At Visit 1, patients will be included after carefully reviewing all inclusion and exclusion criteria. All data concerning the index sting, laboratory parameters like IgE and tryptase levels and skin test results will be recorded as well as the concomitant diseases and medication. Visit 2 will be performed after VIT updosing is finished. At this Visit data concerning the immunotherapy - premedication, preparation, updosing protocol, the outcome of possible large, local reactions and SR and changes in diseases and medication will be recorded. One year after reaching the maintenance dose, Visit 3 will be performed. At this Visit data concerning the maintenance phase like premedication and possible side effects will be recorded as well as the outcome of insect stings.
  Insect Venom: Patients receive insect venom immunotherapy. The frequency of systemic side-effects is recorded and compared between patients under antihypertensive treatment and patients not taking antihypertensive drugs.
Period: Overall Study
Arm/Group | Patients With a History of an Anaphylactic Sting Reaction
Started | 1425 (1425 patients were included in the study (=Visit 1))
Number of Patients Who Performed VIT | 1342 (Visit 2 was performed with 1342 patients)
Completed | 1186 (Visit 3 was performed with 1186 patients)
Not Completed | 239

BASELINE CHARACTERISTICS:
Population: Patients included in the study at Visit 1.
Groups:
- Patients With a History of an Anaphylactic Sting Reaction: At Visit 1, patients will be included after carefully reviewing all inclusion and exclusion criteria. All data concerning the index sting, laboratory parameters like IgE and tryptase levels and skin test results will be recorded as well as the concomitant diseases and medication. Visit 2 will be performed after VIT updosing is finished. At this Visit data concerning the immunotherapy - premedication, preparation, updosing protocol, the outcome of possible large, local reaction and SR and changes in diseases and medication will be recorded. One year after reaching the maintenance dose, Visit 3 will be performed. At this Visit data concerning the maintenance phase like premedication and possible side effects will be recorded as well as the outcome of insect stings.
  Insect Venom: Patients receive insect venom immunotherapy. The frequency of systemic side-effects is recorded and compared between patients under antihypertensive treatment and patients not taking antihypertensive drugs.
Arm/Group | Patients With a History of an Anaphylactic Sting Reaction
Number analyzed (Participants) | 1425
Age, Continuous [Median (Full Range); unit: years] | 52 [35 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 810
  Male | 615
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Side Effects (=Systemic Reaction, SR) During Venom Immunotherapy (VIT)
Description: The primary objective of this study is to evaluate whether subjects under antihypertensive treatment with beta-blockers and/or angiotensin converting enzyme (ACE)-inhibitors show more side effects during VIT compared to subjects with no antihypertensive treatment.
Time Frame: after finishing the updosing phase (duration up to 6 months depending on the updosing protocol chosen by the patient) of a patient's venom immunotherapy; duration of Visit ~1hour
Population: 1342 patients underwent VIT and performed Visit 2. Of these 1342 patients, 93 experienced a systemic side effect during the updosing phase of VIT. Data were missing for 10 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Who Underwent VIT Updosing: Visit 2 will be performed after VIT updosing is finished. At this Visit data concerning the immunotherapy - premedication, preparation, updosing protocol, the outcome of possible large, local reactions and SR and changes in diseases and medication will be recorded.
  The frequency of systemic side-effects is recorded and compared between patients under antihypertensive treatment and patients not taking antihypertensive drugs.
Arm/Group | Patients Who Underwent VIT Updosing
Number analyzed (Participants) | 1332
Participants
  number of patients with SR with AHT treatment: number analyzed (Participants) | 338
  number of patients with SR with AHT treatment | 19
  number of patients with SR without AHT treatment: number analyzed (Participants) | 994
  number of patients with SR without AHT treatment | 74
Statistical Analysis 1: Comparison: Patients Who Underwent VIT Updosing; It was assumed that 24% of the patients would be on β-blockers and/or ACE inhibitors (ACEI). A χ2 test with a two-sided 5% significance level has an 80% power to detect the difference between the group without antihypertensive medication with 6% SR during VIT and the group on β-blockers and/or ACEI with 12.3% SR during VIT (OR = 2.2) when the sample sizes are 631 and 200, respectively. A drop-out rate of 37% was assumed which resulted in a required number of 1,319 patients; Test type: Other — All patients participating in this study belong to one of the following two groups for analysis: the group with antihypertensive treatment (β-blockers or ACEI) and the group without such treatment. The primary outcome was analyzed using logistic linear mixed models with a random intercept. This model type takes into account the clustered structure of the data, i.e., observations clustered in the different participating centers; p = 0.25, Mixed Models Analysis — The level of significance was set at 0.05; Missing at random was assumed, and multiple imputations were conducted with 50 imputations taking into account the cluster design

2. Secondary Outcome: Severity of Sting Reactions
Description: To evaluate whether subjects under antihypertensive treatment with beta-blockers and/or ACE-inhibitors have more severe sting reactions.
Time Frame: duration of first visit (~1hour)
Population: 1425 patients were included in the study at Visit 1. Of these 1425 patients, 603 initially experienced a severe (=Grade 3 and 4 according to the classification of Ring and Messmer), systemic sting reaction. Data were missing for 2 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a History of an Anaphylactic Sting Reaction: At Visit 1, patients will be included after carefully reviewing all inclusion and exclusion criteria. All data concerning the index sting, laboratory parameters like IgE and tryptase levels and skin test results will be recorded as well as the concomitant diseases and medication. The severity of the systemic sting reaction is compared between patients under antihypertensive treatment and patients not taking antihypertensive drugs.
Arm/Group | Patients With a History of an Anaphylactic Sting Reaction
Number analyzed (Participants) | 1423
Participants
  severe reactions in patients with AHT treatment: number analyzed (Participants) | 388
  severe reactions in patients with AHT treatment | 171
  severe reactions in patients without AHT treatment: number analyzed (Participants) | 1035
  severe reactions in patients without AHT treatment | 432
Statistical Analysis 1: Comparison: Patients With a History of an Anaphylactic Sting Reaction; Test type: Other — All patients participating in this study belong to one of the following two groups for analysis: the group with antihypertensive treatment (β-blockers or ACE inhibitors) and the group without such treatment. The secondary outcomes was analyzed using logistic linear mixed models with a random intercept. This model type takes into account the clustered structure of the data, i.e., observations clustered in the different participating centers; p = 0.29, Mixed Models Analysis — The level of significance was set at 0.05; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Correlation of the Prevalence of Cardiovascular Diseases and/or Hypertension With the Risk for More Severe Systemic Sting Reactions.
Description: To correlate the prevalence of cardiovascular diseases and/or hypertension with the risk for more severe systemic sting reactions.
Time Frame: duration of first visit (~1hour)
Population: Correlation cardiovascular disease with risk of more severe systemic sting reaction: 601 of 1425 patients (Visit 1) experienced a severe systemic sting reaction. Datasets missing:9
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Anaphylactic Sting Reaction: At Visit 1, patients will be included after carefully reviewing all inclusion and exclusion criteria. All data concerning the index sting, laboratory parameters like IgE and tryptase levels and skin test results will be recorded as well as the concomitant diseases and medication.
Arm/Group | Patients With Anaphylactic Sting Reaction
Number analyzed (Participants) | 1416
Participants
  severe sting reaction, cardiovascular disease: number analyzed (Participants) | 571
  severe sting reaction, cardiovascular disease | 258
  severe sting reaction, no cardiovascular disease: number analyzed (Participants) | 845
  severe sting reaction, no cardiovascular disease | 343
Statistical Analysis 1: Comparison: Patients With Anaphylactic Sting Reaction; Analysis for correlation of the prevalence of cardiovascular diseases and/or hypertension with the risk for more severe systemic sting reactions; Test type: Other — All patients participating in this study belong to one of the following two groups for analysis: the group with antihypertensive treatment (β-blockers or ACE inhibitor) and the group without such treatment. The secondary outcomes were analyzed using logistic linear mixed models with a random intercept. This model type takes into account the clustered structure of the data, i.e., observations clustered in the different participating centers; p = 0.04, Mixed Models Analysis — The level of significance was set at 0.05. Correlation of the prevalence of cardiovascular diseases and/or hypertension with the risk for more severe systemic sting reactions (p=0.04); [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Association of Bee Venom With a Higher Frequency of Side-effects (=Systemic Reaction, SR).
Description: To evaluate whether bee venom is associated with a higher frequency of side-effects.
Time Frame: as for outcome 1
Population: 1342 patients underwent VIT and performed Visit 2. Of these 1342 patients, 93 experienced a systemic side effect during the updosing phase of VIT. Data missing for 10 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Who Underwent VIT Updosing: Visit 2 will be performed after VIT updosing is finished. At this Visit data concerning the immunotherapy - premedication, preparation, updosing protocol, the outcome of possible large, local reaction and SR and changes in diseases and medication will be recorded.
  The frequency of systemic side-effects is recorded and compared between patients under antihypertensive treatment and patients not taking antihypertensive drugs.
Arm/Group | Patients Who Underwent VIT Updosing
Number analyzed (Participants) | 1332
Participants
  SR in patients treated with bee venom: number analyzed (Participants) | 414
  SR in patients treated with bee venom | 54
  SR in patients treated with vespid venom: number analyzed (Participants) | 918
  SR in patients treated with vespid venom | 39
Statistical Analysis 1: Comparison: Patients Who Underwent VIT Updosing; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.001, Mixed Models Analysis — The level of significance was set at 0.05; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Correlation of High Specific Immunoglobulin E (sIgE) Levels to a Higher Frequency of Side-effects (=Systemic Reaction, SR).
Description: To evaluate whether high specific immunoglobulin E (sIgE) levels are correlated to a higher frequency of side-effects.
  sIgE levels are expressed in kilo units/liter [kU/L].
Time Frame: as for outcome 1
Population: 1342 patients underwent VIT and performed Visit 2. Of these 1342 patients, 93 experienced a systemic side effect during the updosing phase of VIT. sIgE levels were only available for 1009 patients, the other data (=333) are missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Underwent VIT Updosing
Number analyzed (Participants) | 1009
Participants
  SR, bee venom, IgE >0.35-3.5 kU/L: number analyzed (Participants) | 113
  SR, bee venom, IgE >0.35-3.5 kU/L | 17
  SR, bee venom, IgE >3.5-17.5 kU/L: number analyzed (Participants) | 114
  SR, bee venom, IgE >3.5-17.5 kU/L | 17
  SR, bee venom, IgE >17.5 kU/L: number analyzed (Participants) | 53
  SR, bee venom, IgE >17.5 kU/L | 8
  SR, vespid venom, IgE >0.35-3.5 kU/L: number analyzed (Participants) | 287
  SR, vespid venom, IgE >0.35-3.5 kU/L | 17
  SR, vespid venom, IgE >3.5-17.5 kU/L: number analyzed (Participants) | 290
  SR, vespid venom, IgE >3.5-17.5 kU/L | 9
  SR, vespid venom, IgE >17.5 kU/L: number analyzed (Participants) | 152
  SR, vespid venom, IgE >17.5 kU/L | 4
Statistical Analysis 1: Comparison: Patients Who Underwent VIT Updosing; Analysis for sIgE levels - bee venom; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.99, Mixed Models Analysis — The level of significance was set at 0.05; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Patients Who Underwent VIT Updosing; Analysis for sIgE levels - vespid venom; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.15, Mixed Models Analysis — The level of significance was set at 0.05; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Correlation of High Tryptase Levels to a Higher Frequency of Side-effects (=Systemic Reaction, SR).
Description: To evaluate whether high tryptase levels are correlated to a higher frequency of side-effects
Time Frame: as for outcome 1
Population: 1342 patients underwent VIT and performed Visit 2. Of these 1342 patients, 93 experienced a systemic side effect during the updosing phase of VIT. Tryptase levels were only available for 1204 patients. Data missing for 138 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Underwent VIT Updosing
Number analyzed (Participants) | 1204
Participants
  SR in patients with tryptase <11.4µg/L: number analyzed (Participants) | 1084
  SR in patients with tryptase <11.4µg/L | 74
  SR in patients with tryptase >11.4µg/L: number analyzed (Participants) | 120
  SR in patients with tryptase >11.4µg/L | 13
Statistical Analysis 1: Comparison: Patients Who Underwent VIT Updosing; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.16, Mixed Models Analysis — The level of significance was set at 0.05; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Correlation of Quicker Up-dosing Protocols to a Higher Frequency of Side-effects (=Systemic Reaction, SR).
Description: To evaluate whether quicker up-dosing protocols are correlated to a higher frequency of side-effects.
Time Frame: depends on the protocol used for venom immunotherapy, a maximum of about 6 months
Population: 1342 patients underwent VIT and performed Visit 2. Of these 1342 patients, 93 experienced a systemic side effect during the updosing phase of VIT. Data concerning the updosing protocol used were available for 1321 patients; data missing for 21 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Underwent VIT Updosing
Number analyzed (Participants) | 1321
Participants
  SR in patients with conventional updosing: number analyzed (Participants) | 109
  SR in patients with conventional updosing | 5
  SR in patients with quicker updosing: number analyzed (Participants) | 1212
  SR in patients with quicker updosing | 84
Statistical Analysis 1: Comparison: Patients Who Underwent VIT Updosing; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.50, Mixed Models Analysis — The level of significance was set at 0.05; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Efficacy of VIT
Description: The outcome (systemic reaction to sting or not) of sting challenges and/or field stings will be recorded to identify patients who will not tolerate but react to future stings. These results will be compared between patients not taking antihypertensive (AHT) drugs and patients taking AHT drugs.
Time Frame: 1 year after reaching the maintenance dose; duration of Visit ~1hour
Population: Visit 3 was performed with 1186 patients one year after reaching the maintenance phase of VIT. Data missing for 4 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Who Underwent VIT for at Least 1 Year: One year after reaching the maintenance dose, Visit 3 will be performed. At this Visit data concerning the maintenance phase like premedication and possible side effects will be recorded as well as the outcome of insect stings.
  The outcome (systemic reaction or not) of insect stings is recorded and compared between patients under antihypertensive treatment and patients not taking antihypertensive drugs.
Arm/Group | Patients Who Underwent VIT for at Least 1 Year
Number analyzed (Participants) | 1182
Participants
  SR after sting, AHT treatment: number analyzed (Participants) | 296
  SR after sting, AHT treatment | 4
  SR after sting, no AHT treatment: number analyzed (Participants) | 886
  SR after sting, no AHT treatment | 15
Statistical Analysis 1: Comparison: Patients Who Underwent VIT for at Least 1 Year; Test type: Other; p = 0.72, Fisher Exact — The level of significance was set at 0.05

9. Secondary Outcome: Correlation of the Prevalence of Cardiovascular Diseases and/or Hypertension With the Risk for More Frequent Side Effects (=Systemic Reaction, SR) Under VIT.
Description: To correlate the prevalence of cardiovascular diseases and/or hypertension with the risk for more frequent side effects (=systemic reaction, SR) under VIT..
Time Frame: duration of Visit ~1hour
Population: Correlation cardiovascular disease with risk of more frequent side effects under VIT: 93 of 1342 patients (Visit 2) experienced a SR. Datasets missing:17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Underwent VIT Updosing
Number analyzed (Participants) | 1325
Participants
  systemic side-effect, cardiovascular disease: number analyzed (Participants) | 528
  systemic side-effect, cardiovascular disease | 30
  systemic side-effect, no cardiovascular disease: number analyzed (Participants) | 797
  systemic side-effect, no cardiovascular disease | 63
Statistical Analysis 1: Comparison: Patients Who Underwent VIT Updosing; Analysis for correlation of the prevalence of cardiovascular diseases and/or hypertension with the risk for more frequent SR under VIT; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.11, Mixed Models Analysis — The level of significance was set at 0.05; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Not applicable since study is an observational study.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Patients With a History of an Anaphylactic Sting Reaction
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT04269629/Prot_SAP_000.pdf